CLINICAL TRIAL: NCT03758105
Title: Transcranial Direct Current Stimulation (tDCS) Cost-utility-analysis in Medical Care on Depressive Episode With One Drug Therapy Failure.
Acronym: DISCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC17_0493
Record Dates: First submitted 2018-11-23; First posted 2018-11-29 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Depression
Keywords: Depression; psychiatry; health economics; Neurostimulation; tDCS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care and tDCS (Arm A) (Experimental): Arm A patient receives a first tDCS treatment in association with usual care (medication, psychotherapy...). If the patient is responding to tDCS, he can have other tDCS treatments in case of relapse.
  Interventions: Other: tDCS associated with usual care
- Usual care without tDCS (Arm B) (Active Comparator): Arm B patient receives usual care: medication management and psychotherapy.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: tDCS associated with usual care — A tDCS cure will be given to the group "tDCS", one week after their randomization.
  This will be done in association with usual care: medication and psychotherapy Parameters: Anodal stimulation on dorso-lateral prefrontal cortex left, 2mA current.
  Treatment will consist of 15 days with 30 minutes stimulation per day, 5 days a week for 3 weeks.
  Arms: Usual care and tDCS (Arm A)
Other: Usual care — Medication and psychotherapy as prescribed in usual care
  Arms: Usual care without tDCS (Arm B)

SUMMARY:
The purpose of this study is to determine the transcranial direct current stimulation (tDCS) cost-utility in the depression therapy.

This is a 3 years medico-economics study with 1 year follow-up period involving patients with 1 or 2 depression treatment(s) failed.

Eligible subject will be randomized in 2 groups, usual care with tDCS cure (arm A) or only usual care (arm B).

DETAILED DESCRIPTION:
Transcranial direct current stimulation is a non-invasive brain neuromodulation technique. tDCS can be a new therapy in depression.

This study focuses on tDCS cost-utility-analysis. Each patient is following during 12 months. Patients are randomized in 2 arms. Arm A usual care with tDCS cure or arm B usual care without tDCS.

Patient in arm A get a initial tDCS cure one week after randomization. If these patients are answering to the treatment, they can have a new cure in case of relapse. This new cure can start from the second month following initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Depression according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) with 1 or 2 failed antidepressant treatments for the current episode.
* MADRS score superior or equal to 15.
* Patient agreeing to participate in the study
* Patient able to answer questionnaires and able to go at research center for follow-up visit.
* Patient with social insurance

Exclusion Criteria:

* Electroconvulsive therapy or repetitive transcranial magnetic stimulation for current depressive episode.
* Depressive episode with psychotic symptoms or mixed.
* Schizophrenia or addiction to another substance than nicotine
* Severe neurological disorder (like epilepsy, neurological affect, neurological disease)
* Severe and / or progressive somatic pathology (leave to the investigator judgment) preventing from participation in the study.
* tDCS specific contraindications (intracerebral metallic implant, pacemaker)
* Pregnancy or breast feeding.
* Woman of childbearing age without contraception (hormonal or with medical device).
* Participation in another interventional clinical trial
* legal protection
* Persons incarcerated or in obligation of treatment / medical treatment order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-11-11 (Estimated); Study Completion 2023-11-11 (Estimated)

PRIMARY OUTCOMES:
Cost-utility ratio, according to collective perspective of tDCS use in depression compared to usual care without active tDCS. | 12 months
  The utility will be measured by :
  Quality Adjusted Life Year (QALYs) as estimated from responses to the Euroqol-5 Dimensions (EQ-5D) health-related quality of life questionnaire. The questionnaire focuses on 5 dimensions: mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression. For each of these dimensions, 5 answers are possible.
  The costs will be measured by the addition of the following costs:
  Drugs dispensing via Health insurance database "National system of information of the French health insurance" (SNIIRAM), hospitalizations, work stoppages and care consumption collected in a declarative patient questionnaire.

SECONDARY OUTCOMES:
Budget impact analysis of spreading the most efficient strategy for using tDCS | 5 years
  Comparison of intervention costs on the study sample and projection of these costs over 5 years, from the health insurance and hospital perspectives
Response rate | at baseline, at the end of each tDCS cure (for Arm A patients) through study completion (12 months) and at 12 months for all patients
  Response is defined as follows: decrease of the MADRS score by at least 50% compared to baseline score. MADRS stands for Montgomery-Asberg Depression Rating Scale. It is used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. A score from 0 to 6 being normal/symptom absent and a score >34 being severe depression.
Remission rate | 12 months
  Remission rate is defined as follows: MADRS score < 10 (see detailed description of MADRS in outcome 3)
Relapse-free survival | 12 months
  Number of patients with no relapse. Relapse is defined as follows: MADRS ≥ 20 (see detailed description of MADRS in outcome 3)
MADRS score | At Baseline, one month, 2 months, 6 months and 12 months.
  MADRS score (see detailed description of MADRS in outcome 3)
Beck Depression Inventory (BDI) score | At Baseline, one month, 2 months, 6 months and 12 months.
  The BDI is 13-item multiple-choice self-report inventory, for measuring the severity of depression. The global score is an addition of each item's score and ranges from 0 (minimal depression) to 39 (severe depression).
Clinical Global Impression (CGI) score | At Baseline, one month, 2 months, 6 months and 12 months.
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. Each scale is rated from 0 to 7. 0 being the best level and 7 the worst level.
MOCA Score (Montreal Cognitive Assessment) | At Baseline, one month, 2 months, 6 months and 12 months.
  Thirty items assessing multiple cognitive domains are contained in the MoCA: short-term memory (5 points); visuospatial abilities via clock drawing (3 points), and a cube copy task (1 point); executive functioning via an adaptation of Trail Making Test Part B (1 point), phonemic fluency (1 point), and verbal abstraction (2 points); attention, concentration, and working memory via target detection (1 point), serial subtraction (3 points), digits forward (1 point), and digits backward (1 point); language via confrontation naming with low-familiarity animals (3 points), and repetition of complex sentences (2 points); and orientation to time and place (6 points)
Adverse events linked to the medical treatment for depression | 12 months
  Number and types of adverse events linked to the medical treatment for depression
Rate of suicide attempts | 12 months
  number of suicide attempts per patient
Rate of suicides | 12 months
  number of suicides
Treatment(s) switch(es) | At Baseline, one month, 2 months, 6 months and 12 months.
  Number of treatment switches per patient
Treatment(s) dose increase | At Baseline, one month, 2 months, 6 months and 12 months.
  Number of drug(s) dose(s) increases prescribed to the patient
Treatments combination(s) | at Baseline, one month, 2 months, 6 months and 12 months.
  List of drugs (name) prescribed to the patient
Declarative drug compliance via the MARS (Medication Adherence Report Scale) | at baseline and at 12 months
  MARS is the Medication Adherence Report Scale, including 10 questions, the global score ranges from 0 to 10, 0 corresponds to the worst drug compliance and 10 to an excellent drug compliance
Declarative drug compliance via the CRS (Clinician Rating Scale) | at baseline and at 12 months
  CRS is the Clinician Rating Scale , including 7 questions, the global score ranges from 1 to 7, 7 being the worst level of drug compliance.
Total number of tDCS sessions | 12 months
  total number of tDCS sessions per patient
Number of days between the successive tDCS cures | 12 months
  Number of days between end of tDCS cure X and beginning of cure X+1, for each patient
Adverse events linked to tDCS | 12 months
  Number and types of adverse events linked to the tDCS
Compliance with tDCS | 12 months
  number of missed sessions over the number of planned sessions, per patient
Patient acceptability of the tDCS technique: Analog Visual Scale | at the end of the first tDCS cure (up to one month)
  Analog Visual Scale of acceptability of the tDCS completed by the patient, ranging from 0 to 10. 0 being "not acceptable" and 10 being "totally acceptable"
professional status | At baseline
  patient's professional status (active, unemployed, retired...)
Impact of the implementation of the tDCS on the organization of care | 12 months
  The organizational impact of the tDCS will be evaluated from the point of view of doctors, nurse and patients: staff, equipment, maintenance, location and mobilization time of these resources, using a specific questionnaire

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU d'Angers, Angers
  - Clinique Mirambeau, Anglet
  - CHRU de Besançon, Besançon
  - Chu Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - Chu de Lyon, Lyon
  - Nantes University Hospital, Nantes
  - Aphp Hopital Saint Antoine, Paris
  - CH Henri Laborit (Poitiers), Poitiers
  - Centre hospitalier Guillaume Regnier Rennes, Rennes
  - CH du Rouvray - Rouen, Rouen
  - CHU de Tours / CHRU de Tours, Tours

REFERENCES:
- [Derived] Sauvaget A, Lagalice L, Schirr-Bonnans S, Volteau C, Pere M, Dert C, Rivalland A, Tessier F, Lepage A, Tostivint A, Deschamps T, Thomas-Ollivier V, Robin A, Pineau N, Cabelguen C, Bukowski N, Guitteny M, Beslot A, Simons L, Network H, Vanelle JM, D'Urso G, Bulteau S, Riche VP; DISCO investigators group. Cost-utility analysis of transcranial direct current stimulation (tDCS) in non-treatment-resistant depression: the DISCO randomised controlled study protocol. BMJ Open. 2020 Jan 13;10(1):e033376. doi: 10.1136/bmjopen-2019-033376. PMID 31937653